CLINICAL TRIAL: NCT06811259
Title: The Effect of Virtual Reality on Pain and Anxiety During Colposcopic Biopsy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ahu AKSOY, Asst. Prof, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 002
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-01

CONDITIONS: Pain and Anxiety
Keywords: Colposcopy, biopsy, virtual reality, anxiety and pain, nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (VR) group (Experimental): For the women in the experimental group, new protective covers will be placed on the headset parts of the VR glasses that the researchers already have before the application. Videos with forest and sea views will be presented to the woman's preference via the VR program loaded onto the phone, the video selected by the woman will be opened and the phone will be inserted into the virtual reality glasses. After the woman is positioned for the gynecological surgical procedure, the virtual reality glasses will be put on and will remain on throughout the procedure. The virtual reality application will be terminated after the colposcopic biopsyis completed. The Visual Analog Scale (VAS) will be filled in during the procedure and 15 minutes after the colposcopic biopsy, and the State-Trait Anxiety Inventory (STAI-S) will be filled in before the colposcopic biopsyand 15 minutes after the colposcopic biopsy.
  Interventions: Other: Virtual reality (in experimental group)
- Control group (Other): Women in the control group will receive only standard care during colposcopic biopsy. The Visual Analog Scale (VAS) will be completed during the procedure and 15 minutes after the colposcopic biopsy, and the State-Trait Anxiety Inventory (STAI-S) will be completed before and 15 minutes after the colposcopic biopsy.
  Interventions: Other: Standart care

INTERVENTIONS:
Other: Virtual reality (in experimental group) — Virtual reality application is performed with virtual reality glasses. Virtual reality glasses are a simulation model that provides participants with the opportunity to communicate with a dynamic environment created by computers and gives them a sense of reality. Virtual reality glasses, which have a mechanism compatible with smart phones, allow videos downloaded to mobile phones or watched directly via the internet to be viewed at a 360-degree angle. The two lenses on the device provide panoramic viewing by dividing the image into two equal parts. The bands on the front of the device that fits the face are flexible and prevent the device from slipping from the face. The buckles on the back are adjustable and provide ease of use. Thanks to the proximity sensor on the device, images can be zoomed in and out to obtain a clearer image. Thanks to the device holder on the sides, the phone can be easily placed and removed from the device. Again, videos can be advanced or changed with the tou
  Arms: Experimental (VR) group
Other: Standart care — Women in the control group will receive only standard care during colposcopy
  Arms: Control group

SUMMARY:
The study was planned as a prospective, two-arm (1:1) randomized controlled experimental study to determine the effect of virtual reality applied during colposcopic biopsy on pain and anxiety. The research hypothesis of the research are as follows; H1a: There is a difference between the pain levels of the virtual reality group and the control group after colposcopic biopsy.

H1b: There is a difference between the anxiety levels of the virtual reality group and the control group after colposcopic biopsy.

DETAILED DESCRIPTION:
Methods: In the study, 82 women who underwent colposcopic biopsy at Mersin University Hospital Gynecological Oncology Polyclinic were randomly assigned to experimental and control groups. Before the application, new protective covers will be attached to the headset parts of the virtual reality (VR) glasses that the researchers already have for each woman in the experimental group. Videos with forest and sea views will be presented to the woman's preference through the VR program loaded on the phone, the video selected by the woman will be opened and the phone will be inserted into the VR glasses. After the woman is positioned for the gynecological surgical procedure, the VR glasses will be put on and will remain on during the procedure. The VR application will be terminated after the colposcopic biopsy is completed. The Visual Analog Scale (VAS) will be filled in during the procedure and 15 minutes after the colposcopic biopsy, and the State-Trait Anxiety Inventory (STAI-S) will be filled in before and 15 minutes after the colposcopic biopsy. Only standard care will be given to women in the control group during colposcopy. The primary expected outcome of the study is the effect of virtual reality on pain in women undergoing colposcopic biopsy. The secondary expected outcome of the study is to determine the effect of virtual reality on anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18,
* Subjected to colposcopic biopsy,
* Not using a medication that directly affects vital signs,
* Not using antidepressants, anxiolytics or sedatives,
* Not using analgesics or anesthetics 24 hours before the procedure,
* Not having any psychiatric illness,
* Not having vision, hearing or perception problems,
* Not having communication problems (can speak Turkish),
* Women who agree to participate in the study verbally and in writing.

Exclusion Criteria:

* Women under the age of 18,
* Those who have not undergone colposcopic biopsy,
* Those who are taking a medication that directly affects vital signs,
* Those who are taking antidepressants, anxiolytics and sedatives,
* Those who are taking analgesics or anesthetics 24 hours before the procedure,
* Those who have any psychiatric illness,
* Those who have vision, hearing and perception problems,
* Those who have communication problems (cannot speak Turkish),
* Those who have diseases that cause movement sensitivity,
* Those who cannot watch the entire video,
* Women who do not accept to participate in the research verbally or in writing.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Just female
Enrollment: 60 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | change from during the intervention, at the end of 15 minutes
  Visual Analog Scale (VAS) The Visual Analog Scale is used to measure the pain perceived by the person. The individual can indicate their own pain by drawing a line, putting a dot or pointing between the 10 cm (100 mm) section of the scale where there is no pain (zero) on one end and the most severe pain (10) on the other end. The distance from the point where there is no pain to the point marked by the individual is measured in centimeters and the value found indicates the individual's pain intensity. On the VAS scale, 0-44 mm indicates mild pain, 45-74 mm indicates moderate pain, while 75-100 mm reflects severe pain.

SECONDARY OUTCOMES:
Anxiety Assessment | change from before the intervention, at the end of 15 minutes
  State Anxiety Inventory (STAI-S) Anxiety level of women will be evaluated that the "State Anxiety Inventory". The scale consists of 20 items that determine how an individual feels at a certain moment. The items in the four-point Likert-type scale range from 1-4 points (not at all-completely) according to the intensity of the emotions expressed. 10 items in the scale are reverse scored. The lowest score that can be obtained from the scale is "20" and the highest score is "80". The state anxiety score is calculated by adding 50 points to the difference between the total weighted scores of direct and reverse statements. In the evaluation of the scale, the cut-off score was determined as 40. Accordingly, those who score below 40 are considered not to have anxiety, while those who score above 40 are considered to have anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmid BC, Marsland D, Jacobs E, Rezniczek GA. A Preparatory Virtual Reality Experience Reduces Anxiety before Surgery in Gynecologic Oncology Patients: A Randomized Controlled Trial. Cancers (Basel). 2024 May 17;16(10):1913. doi: 10.3390/cancers16101913. PMID 38791991
- [Result] Oz T, Demirci N. The Effect of Virtual Reality, Music Therapy, and Stress Ball Application on Pain and Anxiety During Outpatient Gynecological Procedures: A Randomized Controlled Trial. J Perianesth Nurs. 2024 Dec;39(6):1034-1041. doi: 10.1016/j.jopan.2024.01.022. Epub 2024 May 25. PMID 38795085